CLINICAL TRIAL: NCT00002816
Title: EXTRAMEDULLARY RELAPSE AND OCCULT BONE MARROW INVOLVEMENT IN CHILDHOOD ACUTE LYMPHOBLASTIC LEUKEMIA: A PHASE III GROUP-WIDE STUDY
Brief Title: Combination Chemotherapy in Treating Children With Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1951; CCG-1951 (Other: Children's Cancer Group); CDR0000064968 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-06-23 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; Dexamethasone; Calcium Dobesilate; Etoposide; Idarubicin; Ifosfamide; Leucovorin; Mesna; pegaspargase; Hydrocortisone; Thioguanine; Vincristine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EARLY # CNS RELAPSE with BM DONOR (Experimental): Induction (Etoposide, Ifosfamide with Mesna Uroprotection,Ifosfamide, Dexamethasone, Vincristine sulfate, PEG, ITT (methotrexate, cytosine arabinoside and therapeutic hydrocortisone), and leucovorin calcium then Intensification (4 courses of 6 weeks, ITT, dexamethasone, vincristine, methotrexate, leucovorin, 6-Thioguanine, cytarabine (Ara-C), Etoposide, pegaspargase, Ifosfamide with Mesna) and Idarubicin and CXRT.
  Interventions: Drug: cytarabine; Drug: dexamethasone; Drug: etoposide; Drug: idarubicin; Drug: ifosfamide; Drug: leucovorin calcium; Drug: mesna; Drug: pegaspargase; Drug: therapeutic hydrocortisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Drug: Methotrexate
- LATE CNS RELAPSE with/without BM DONOR, TESTICULAR or OCULAR (Experimental): Induction (Etoposide, Ifosfamide with Mesna Uroprotection,Ifosfamide, Dexamethasone, Vincristine sulfate, pegaspargase, ITT (methotrexate, cytosine arabinoside and therapeutic hydrocortisone), and leucovorin calcium then Intensification (4 courses of 6 weeks, ITT, dexamethasone, vincristine, methotrexate, leucovorin, 6-Thioguanine, cytarabine (Ara-C), Etoposide, PEG, Ifosfamide with Mesna) and Idarubicin), and Maintenance (4 x 12 courses) of ITT, Vincristine, Methotrexate, T-thioguanine.
  Interventions: Drug: cytarabine; Drug: dexamethasone; Drug: etoposide; Drug: idarubicin; Drug: ifosfamide; Drug: leucovorin calcium; Drug: mesna; Drug: pegaspargase; Drug: therapeutic hydrocortisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Drug: Methotrexate

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar-U; NSC-63878
Drug: dexamethasone — Given IV
  Other Names: Decadron; NSC- 34521
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; NSC-14154p
Drug: idarubicin — Given IV
  Other Names: Idamycin; NSC-256439
Drug: ifosfamide — Given IV
  Other Names: Ifex; NSC-109724
Drug: leucovorin calcium
Drug: mesna — Given IV
  Other Names: Mesnex; NSC-113891
Drug: pegaspargase — Given IV
  Other Names: PEG Asparaginase; PEG-ASP; K/H; KYOWA; HAKKO; NSC-644954
Drug: therapeutic hydrocortisone
Drug: thioguanine
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; NSC-675574
Radiation: low-LET cobalt-60 gamma ray therapy
  Arms: LATE CNS RELAPSE with/without BM DONOR, TESTICULAR or OCULAR
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy
Drug: Methotrexate — Given IV
  Other Names: MTX; NSC-740

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase III trial to compare the effectiveness of combination chemotherapy in treating children who have relapsed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Improve the outcome in children with first isolated central nervous system (CNS), testicular, or ocular relapse of acute lymphoblastic lymphoma (ALL), and increase the knowledge of the characteristics of extramedullary and subsequent relapses of ALL. II. Quantitate, by current molecular biologic techniques, occult systemic leukemia in cases of conventional isolated extramedullary relapse, and examine the relationship between this assessment and subsequent clinical outcome, particularly overt marrow relapse. III. Quantitate occult systemic leukemia in subsets of extramedullary relapse that include site (CNS, testis, or eye), time of relapse (early or late), initial risk group, immunophenotype, DNA index and karyotype, gender (for CNS and eye), and ethnicity, and assess the response to therapy in patients entered on companion protocol CCG-B958. IV. Compare the relative sensitivities of two quantitative in vitro assays for occult systemic leukemia (fluorescence-activated cell sorter/leukemic progenitor cell clonogenic assay vs. polymerase chain reaction-based clonospecific assay), correlate the assays with clinical outcome, and assess other biologic studies of leukemic cells (e.g., neurotropic potential in the SCID mouse xenograft model and methotrexate sensitivity). V. Determine the event-free survival (EFS) and pattern of failure in children with first isolated CNS, testicular, or ocular relapse after treatment that includes intensive systemic chemotherapy. VI. Correlate EFS in patients with CNS and ocular relapse with sex, and in patients with relapse at all three sites with ethnicity. VII. Evaluate the impact of combined chemotherapy and radiotherapy on health status in survivors at two and four years after extramedullary relapse and study entry.

OUTLINE: All patients receive induction chemotherapy over 5 weeks with: etoposide, ifosfamide/mesna, dexamethasone, vincristine, and pegaspargase (if pegaspargase is not available, E. coli asparaginase may be substituted throughout study); then dexamethasone, vincristine, pegaspargase (or E. coli asparaginase), and high-dose methotrexate with leucovorin rescue; and triple intrathecal chemotherapy (TIT). Following induction chemotherapy, all patients receive two 6-week courses of intensification therapy with intermittent TIT; each course consists of dexamethasone, vincristine, high-dose methotrexate/leucovorin, thioguanine, cytarabine, etoposide, and pegaspargase (or E. coli asparaginase) followed by dexamethasone, vincristine, high-dose methotrexate/leucovorin, thioguanine, ifosfamide/mesna, and idarubicin. Patients receive 2 additional courses of intensification chemotherapy followed by four 12-week courses of maintenance chemotherapy with vincristine and methotrexate every 2 weeks and daily oral thioguanine. Total duration of therapy is 78 weeks. Patients with isolated ocular relapse receive local radiotherapy prior to initiation of induction chemotherapy; those who also have CNS leukemia begin TIT with the radiotherapy. Patients with CNS relapse receive craniospinal irradiation during the first month of maintenance therapy, with the dose and fields based on whether they will receive TBI and whether they have had CNS irradiation previously. Patients with testicular relapse receive bilateral testicular irradiation during the first 3 weeks of intensification therapy. Patients are followed every 3 months for 3 years, every 6 months for 3 years, and yearly thereafter, or upon relapse, second malignancy, loss to follow up, or death. All patients undergo quality-of-life assessment at entry and 2 and 4 years after entry.

PROJECTED ACCRUAL: Approximately 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute lymphoblastic leukemia (ALL) with isolated extramedullary relapse Relapse occurred during or following front-line therapy for ALL Initial diagnosis of more than 25% blasts of L1 or L2 morphology No leukemic marrow (M1) by conventional assessment Patients with B precursor ALL must also be enrolled on study CCG-B958 Relapse occurred in the CNS, testis, or eye Ocular relapse confirmed by an ophthalmologist and by cytology or iris biopsy Combined CNS and ocular relapse eligible Down Syndrome patients not eligible No prior bone marrow transplantation in first remission No prior toxicity from any study drugs Patient age: Under 21

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 1996-12; Primary Completion 2002-11 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Event Free Survival
  The evaluation of the relationship between prognostic or treatment factors and EFS

CONTACTS AND LOCATIONS:
Overall Officials: Michael L.N. Willoughby, MD, Study Chair — Princess Margaret Hospital for Children
Locations (33):
- United States (30):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Result] Uckun FM, Gaynon PS, Stram DO, Sensel MG, Sarquis MB, Willoughby M. Bone marrow leukemic progenitor cell content in pediatric T-lineage acute lymphoblastic leukemia patients with an isolated extramedullary first relapse. Leuk Lymphoma. 2001 Jan;40(3-4):279-85. doi: 10.3109/10428190109057926. PMID 11426549
- [Result] Uckun FM, Gaynon PS, Stram DO, Sensel MG, Sarquis MB, Lazarus KH, Willoughby M. Paucity of leukemic progenitor cells in the bone marrow of pediatric B-lineage acute lymphoblastic leukemia patients with an isolated extramedullary first relapse. Clin Cancer Res. 1999 Sep;5(9):2415-20. PMID 10499612